CLINICAL TRIAL: NCT02506426
Title: Endoscopic Sinus Surgery for Refractory Chronic Sinusitis: A Randomized, Double-blind Controlled Trial
Brief Title: Endoscopic Sinus Surgery for Refractory Chronic Sinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Luke Rudmik, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB15-0809
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Sinusitis
Keywords: Chronic Sinusitis; Chronic Rhinosinusitis; Endoscopic sinus surgery; Septoplasty
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Sinus Surgery + Septoplasty (Active Comparator): A surgery that uses special telescopes through the nostrils to make the nasal septum straight and open the facial sinuses without any incisions. The sinuses are opened using special microscopic instruments and the procedure takes approximately 90 - 120 minutes.
  Interventions: Procedure: Endoscopic sinus surgery + Septoplasty
- Septoplasty alone (Experimental): A surgery that is performed to straighten a bent nasal septum. It is shorter (take approximately 25 - 30 minutes) and less invasive (do not open the facial sinuses) that might provide the same benefits compared to the larger and longer endoscopic sinus surgery.
  Interventions: Procedure: Septoplasty alone

INTERVENTIONS:
Procedure: Endoscopic sinus surgery + Septoplasty — Opening of the paranasal sinuses along with correcting the nasal septum
  Arms: Endoscopic Sinus Surgery + Septoplasty
Procedure: Septoplasty alone — Straightening of the nasal septum without opening the paranasal sinuses
  Arms: Septoplasty alone

SUMMARY:
Chronic sinusitis is a disease involving severe swelling of your facial sinuses and nasal cavity. Chronic sinusitis is a common disorder and roughly 5% of adult men and women have chronic sinusitis in Canada. Surgery has shown to have benefits for people suffering from chronic sinusitis. There are two surgeries which have been shown to help people: 1) Endoscopic sinus surgery with septoplasty and 2) Septoplasty alone. Both surgeries have research which show they help improve quality of life and reduce symptoms. However, it is unknown which surgery is better.

'Endoscopic sinus surgery with Septoplasty' uses special telescopes through the nostrils to make the nasal septum straight and open the facial sinuses without any incisions. The sinuses are opened using special microscopic instruments and the procedure takes approximately 90-120 minutes.

'Septoplasty alone' is a shorter (take approximately 25-30 minutes) and less invasive (do not open the facial sinuses) that might provide the same benefits compared to the larger and longer endoscopic sinus surgery.

Currently, performing 'Endoscopic Sinus Surgery and Septoplasty' together is the standard of care, however, there is limited evidence to support just performing 'Septoplasty alone' provides similar results but it is shorter and has lower risks. This represents a significant gap in the investigators' knowledge, which adversely impacts a doctor's ability to counsel patients who have chronic sinusitis and elect to undergo surgery.

The purpose of this study is to understand which surgery (endoscopic sinus surgery plus septoplasty OR septoplasty alone) is the most appropriate for people with chronic sinusitis. You are being asked to participate in this study because you have chronic sinusitis and are also going to have surgery to improve your quality of life.

DETAILED DESCRIPTION:
Chronic sinusitis, officially known as chronic rhinosinusitis (CRS), is a common yet under-recognized chronic inflammatory disease of the paranasal sinuses affecting approximately 5% of the Canadian population. Aside from gaining a reputation for its detrimental effects on patient quality-of-life (QoL) and daily productivity, CRS is associated with a lifetime of medical and surgical resource consumption resulting in significant health care expenditure. The estimated direct cost of CRS to the Canadian health care system is $990 million per year, which is comparable to the annual direct costs of asthma. The large economic burden of chronic sinusitis provides a strong incentive to improve both the quality and value of care for this chronic inflammatory disease.

Although the etiology of CRS is considered multi-factorial without one single unifying factor, several studies have investigated the role of a septal deviation as a predisposing factor of CRS. A systematic review and meta-analysis quantified the outcomes and concluded that there was statistical evidence for the association between CRS and septal deviation, especially those with a septal deviation angle > 10-degrees. However, the clinical relevance of septal deviation as an etiologic factor for CRS is still unknown.

Based on several recent evidence-based guidelines, sinonasal 'surgery' can be considered for patients with medically refractory CRS as defined by having persistent symptoms despite a minimum of 3 months with topical sinonasal corticosteroid therapy along with a minimum of a 7-day course of systemic corticosteroid +/- 2-week course of broad-spectrum antibiotic. The important question remains, what is the most appropriate surgical intervention for patients with refractory CRS? Currently there are two surgical options for CRS and both procedures have non-randomized evidence to support their beneficial effects in this patient population: (1) Septoplasty alone (ie. only correcting the deviated septum and not dissecting into the paranasal sinuses), and (2) Endoscopic sinus surgery (ESS) along with a septoplasty (ie. correcting the septal deviation and opening up the paranasal sinuses). With an estimated direct health care cost exceeding $100 million spent on sinonasal surgery in Canada for management of CRS, optimizing the allocation of scarce surgical resources toward interventions with the most proven benefit would result in significant improvements in both the quality and value of care to patients.

In 2005, a prospective non-randomized study compared septoplasty alone to septoplasty plus ESS. They demonstrated that septoplasty alone had a 93% subjective success rate for patients with CRS which was no different than the 88% success rate of ESS plus septoplasty. Although this study has provided some insight into this topic, it was limited by the lack of randomization, lack of stringent inclusion criteria for refractory CRS, and lack of using a validated patient-reported outcome measure. Since 2004, there have been several prospective observational cohort studies evaluating the role of ESS in patients with refractory CRS. Overall the outcomes from these studies suggest that ESS provides improved patient-reported outcomes and objective outcomes. However, despite excellent observational evidence supporting both septoplasty and ESS, there has never been a robust randomized controlled trial (RCT) to prove additional benefit of ESS compared to septoplasty alone for patients with CRS.

In real world practice, ESS is commonly performed in combination with septoplasty despite the lack of a RCT. The lack of level-1 evidence continues to raise questions regarding the true effectiveness and appropriateness of ESS for patients with CRS as opposed to just performing a septoplasty alone. This current gap in the literature provides a strong incentive to evaluate the role of ESS using a RCT design and is the impetus behind this research project.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of CRS WITHOUT nasal polyps (as per Canadian Rhinosinusitis Guidelines22)
3. Septal deviation greater then 10-degrees on the CT sinuses scan10.
4. Failed medical therapy as defined by having persistent symptoms and reduced disease-specific QoL despite receiving a minimum of the following treatment: 3 months topical sinonasal corticosteroid therapy along with a minimum of a 7-day course of systemic corticosteroid + 2-week course of broad-spectrum antibiotic13.
5. Lund-MacKay CT Sinus score ≥ 5 points23.
6. Patient elects to proceed with a surgical intervention for their medically refractory CRS.
7. Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study.
8. Participants must sign an informed consent document indicating that they understand the purpose of and procedures of the study and are willing to participate in the study

Exclusion Criteria:

1. Women who are pregnant or breast feeding or plan to become pregnant during the study period.
2. History of prior sinus or septal surgery.
3. Participants who will not be able to complete the follow-up appointments/evaluations.
4. Have significant oral structural abnormalities, eg. Un-repaired cleft palate.
5. History of a systemic inflammatory disease (eg. Sarcoidosis), primary ciliary dyskinesia, or systemic vasculitis (eg. granulomatosis with polyangiitis (GPA)).
6. Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the participant's participation or compliance with the study.
7. Inability to read and understand English.
8. Any participant who unfit to undergo surgery under general anesthesia .
9. Current participation in another clinical trial at the time of the screening visit.
10. Any patient that the investigator has reason to believe that they will not follow the study procedures, treatment and/or follow-up schedule.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Disease specific-quality of life using the 22-item sinonasal outcome test (SNOT-22) | Change in baseline compared to 12 months post surgery
  The SNOT-22 is validated quality of life (QoL) questionnaire and it is 22-item outcome measure applicable to both sinonasal conditions and surgical treatments (score range: 0-110). Derived from the SNOT-20, two additional questions were added to measure nasal blockage and sense of taste/smell. Lower total scores on the SNOT-22 imply better QoL.

SECONDARY OUTCOMES:
Strength of Patient Blinding using a group selection scale | 3 months after surgery
  Will ask patients to select one of the following options regarding what they feel is their treatment group: a) Septoplasty alone group, b) ESS + Septoplasty group, or c) Don't know.
Generic quality of life using the EQ-5D questionnaire | Change in baseline compared to 12 months post surgery
  It is a generic health state utility metric which contains five attributes: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression.
Daily productivity using the Work Productivity and Activity Impairment (WPAI) questionnaire | Change in baseline compared to 12 months post surgery
  Assesses the work productivity losses from being in a certain health state.
Adherence/compliance to medical therapy using the Morisky 8-item Adherence Questionnaire | Change in baseline compared to 12 months post surgery
  Measures the compliance to medical therapy prescribed after surgery
Patient Satisfaction with care using the Patient Satisfaction Questionnaire Short-form (PSQ-18) | Change in baseline compared to 12 months post surgery
  Measures patient satisfaction with the therapy they have received

CONTACTS AND LOCATIONS:
Overall Officials: Candice Werner, Study Director — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Ottawa, Ottawa, Ontario